CLINICAL TRIAL: NCT00005576
Title: A PHASE I STUDY OF CHIMERIC HUMAN/MURINE ANTI-GD2 MONOCLONAL ANTIBODY (ch14.18) WITH GM-CSF AND INTERLEUKIN-2 (IL-2) IN CHILDREN WITH NEUROBLASTOMA IMMEDIATELY POST AUTOLOGOUS BMT OR PBSC RESCUE
Brief Title: Monoclonal Antibody Therapy With Sargramostim and Interleukin-2 in Treating Children With Neuroblastoma
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2012-01527; 0935; CDR0000063533 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2000-05-02; First posted 2003-11-05 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Disseminated Neuroblastoma; Recurrent Neuroblastoma; Regional Neuroblastoma
MeSH Terms: conditions — Neuroblastoma | interventions — dinutuximab; Isotretinoin; aldesleukin; Interleukin-2; sargramostim; Granulocyte-Macrophage Colony-Stimulating Factor

ARMS (1):
- Treatment (monoclonal antibody Ch14.18, aldesleukin) (Experimental): Patients receive MOAB IV over 5 hours on days 7-10 during courses 2 and 4 and on days 3-6 during courses 1, 3, and 5; sargramostim (GM-CSF) IV over 2 hours or subcutaneously daily on days 0-13 during courses 1, 3, and 5; interleukin-2 IV continuously on days 0-3 and 7-10 during courses 2 and 4; and oral isotretinoin twice daily on days 14-27 during courses 2 and 4 and on days 10-23 during courses 3 and 5. Treatment repeats every 24-32 days for 5 courses in the absence of unacceptable toxicity.
  Interventions: Biological: monoclonal antibody Ch14.18; Drug: isotretinoin; Biological: aldesleukin; Biological: sargramostim

INTERVENTIONS:
Biological: monoclonal antibody Ch14.18 — Given IV
  Other Names: Ch14.18; MOAB Ch14.18
Drug: isotretinoin — Given orally
  Other Names: 13-CRA; Amnesteem; Cistane; Claravis; Sotret
Biological: aldesleukin — Given IV
  Other Names: IL-2; Proleukin; recombinant human interleukin-2; recombinant interleukin-2
Biological: sargramostim — Given IV
  Other Names: GM-CSF; Leukine; Prokine

SUMMARY:
Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Colony-stimulating factors such as sargramostim may increase the number of immune cells found in bone marrow or peripheral blood. Interleukin-2 may stimulate a person's white blood cells to kill cancer cells. Combining monoclonal antibody therapy with sargramostim or interleukin-2 may kill more tumor cells. Phase I trial to study the effectiveness of monoclonal antibody therapy given with sargramostim and interleukin-2 in treating children with neuroblastoma who have just completed bone marrow or peripheral stem cell transplantation

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Determine the maximum tolerated dose of monoclonal antibody (MOAB) ch14.18 when combined with sargramostim (GM-CSF) and interleukin-2 (IL-2) after autologous bone marrow or peripheral blood stem cell rescue in children with neuroblastoma.

II. Determine the toxic effects of this regimen in these patients. III. Determine the pharmacokinetics, including antibody level, antibody-binding activity, and presence of human anti-chimeric antibodies, of this regimen in these patients.

IV. Determine the activity of IL-2 and MOAB ch14.18 against tumor cells in terms of response using standard clinical measurements such as bone marrow immunocytology in these patients.

V. Determine the extent of coating of tumor cells (bone marrow metastases) by MOAB ch14.18 in these patients.

VI. Determine the feasibility of isotretinoin administered between courses beginning after course 2 in these patients.

OUTLINE: This is a multicenter, dose-escalation study of monoclonal antibody (MOAB).

Patients receive MOAB IV over 5 hours on days 7-10 during courses 2 and 4 and on days 3-6 during courses 1, 3, and 5; sargramostim (GM-CSF) IV over 2 hours or subcutaneously daily on days 0-13 during courses 1, 3, and 5; interleukin-2 IV continuously on days 0-3 and 7-10 during courses 2 and 4; and oral isotretinoin twice daily on days 14-27 during courses 2 and 4 and on days 10-23 during courses 3 and 5. Treatment repeats every 24-32 days for 5 courses in the absence of unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of MOAB until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity. A minimum of 6 additional patients are treated at the MTD.

Patients are followed every other week for 2 months and then every 3 months for 6 months.

PROJECTED ACCRUAL: Approximately 6-16 patients will be accrued for this study within 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Must have recently completed a course of myeloablative therapy followed by autologous stem cell (bone marrow or peripheral blood) rescue (ASCT)
* Patients must have a diagnosis of neuroblastoma based upon tumor histology or bone marrow metastases and elevated urine catecholamine metabolites; greater than 98% of neuroblastomas are GD2-positive without intratumor heterogeneity, so these tumors will not be immunostained prior to study entry
* Patients entered on CCG-3951 may become eligible following the third course of high-dose chemotherapy followed by peripheral blood stem cell (PBSC) rescue; patients treated on institutional (local) protocols of high-dose chemotherapy with PBSC rescue may also become eligible after one or more courses of PBSC rescue
* Patients must enter onto study within 8 weeks after the total absolute phagocyte count [neutrophils (segs + bands) + monocytes] is > 1,000/uL; the APC criteria include counts obtained while on G-CSF therapy
* Patients must have a performance status of 0, 1 or 2 and patients must have a life expectancy of >= 2 months
* Serum creatinine =< 1.5 x normal, or creatinine clearance or radioisotope glomerular filtration rate (GFR) >= 60 ml/min/1.73 m^2
* Total bilirubin =< 1.5 x normal
* Serum glutamic oxaloacetic transaminase (SGOT) (aspartate aminotransferase [AST]) or serum glutamate pyruvate transaminase (SGPT) (alanine aminotransferase [ALT]) =< 5 x normal
* Veno-occlusive disease, if present, should be stable or improving
* Shortening fraction of >= 27% by echocardiogram, or ejection fraction of > 50% by gated radionuclide study
* Forced expiratory volume in 1 second (FEV1) and forced vital capacity (FVC) > 60% of predicted by pulmonary function test
* For children who are unable to do pulmonary function tests (PFTs), no evidence of dyspnea at rest, no exercise intolerance, and a pulse oximetry > 94% on room air
* Patients with seizure disorder may be enrolled if on anticonvulsants and well controlled
* Central nervous system (CNS) toxicity < grade 2
* Patients must have a double lumen catheter or single lumen and peripheral IV so that interleukin (IL)-2 and ch14.18 can be given separately
* Patients who remain evaluable for response on Phase II/III studies (i.e. CCG-3891) are not eligible for this study; however, patients treated on Phase I studies (i.e. CCG-3951) and patients who are no longer evaluable on Phase II/III studies (i.e. progressive disease following therapy) will be eligible
* Patients who were previously treated with antibody 14.G2a or ch14.18 are ineligible for this study
* Patients requiring chronic use of corticosteroids are ineligible
* Corticosteroid, immunosuppressive drugs, myelosuppressive chemotherapy, and retinoic acid must not be given within 14 days prior to study entry
* Radiation therapy must not be given within seven days prior to study entry or during therapy
* All patients and/or their parents or legal guardians must sign a written informed consent
* All institutional, FDA, and NCI requirements for human studies must be met

Max Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 6 (Actual)
Dates: Start 2001-01; Primary Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose of monoclonal antibody (MOAB) ch14.18 when combined with sargramostim and IL-2 after autologous bone marrow or peripheral blood stem cell rescue in children with neuroblastoma | 32 days

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Gilman, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Arcadia, California, United States